CLINICAL TRIAL: NCT01487213
Title: Routine Follow-up Versus Self-assessment of Complete Abortion Following Medical Abortion, Effect on Its Success and Acceptability: a Randomized Controlled Trial
Brief Title: Routine Follow-up Versus Self-assessment in Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ullevaal University Hospital (Other); University of Helsinki (Other); Gynmed Clinic Vienna (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, professor, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WNI1000
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Medical Abortion
Keywords: Medical abortion; Termination of pregnancy; Mifepristone; Misoprostol; Urine hCG; Follow Up; Termination of unwanted pregnancy. Self assessment (follow up) after medical abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controls (No Intervention): Routine follow-up at the clinic 2-3 weeks after the treatment
- Home self test (Other): Intervention
  Interventions: Other: Home self assessment of complete medical abortion

INTERVENTIONS:
Other: Home self assessment of complete medical abortion — Self assessment of complete abortion using a home semiquantitative U-hCG test. Follow-up out patient review two-three weeks later by qualified practitioner to evaluate success of procedure using the clinic's standard routine. The patient charts will be reviewed after three months in order to control for possible extra visits related to abortion-related complications.
  Arms: Home self test

SUMMARY:
The main objective of the study is to optimize the routines for follow-up after medical abortion in order to give women more autonomy by reducing the number of consultations involved and to reduce the frequency of postabortal curettage.

This will be achieved by providing means for women for postabortal self-assessment with the use of a quantitative urinary hCG test.

ELIGIBILITY:
Inclusion Criteria:

* women requesting termination of pregnancy by means of mifepristone followed by home administration of misoprostol at < /=63 days of gestation, with no contraindication to medical abortion and self administration of misoprostol at home, and who have given their informed consent will be eligible for study recruitment.

Exclusion Criteria:

* women who do not wish to participate
* women who do not want home administration of misoprostol
* women who are unable to communicate in Swedish, Norwegian, English, Finnish or German and women with symptoms and signs of ectopic pregnancy
* minors (i.e. women < 18 years of age) will not be enrolled for the study.
* women seeking termination of pregnancy with no sign of a visible intrauterine pregnancy (i.e. visible intrauterine yolk sac).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of complete abortions | Until 3 months post treatment
  The primary objective is thus to demonstrate the non-inferiority of self-assessment of complete abortion following medical abortion compared to routine follow-up in terms of the percentage of women requiring surgical abortion, within a margin of non-inferiority of 5%.

SECONDARY OUTCOMES:
postabortion contraception | until 12 months post treatment
  The use of contraception and rate of repeat abortion at follow-up questionnaire at one year.
adverse events | util 3 months post treatment
  Number of women reporting adverse events and side effects including infections, bleeding, pain

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell-Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- GynMed Clinic, Vienna, Austria
- Dept. Obstetrics and Gynaecology,Helsinki University Central Hospital, Helsinki, Finland
- Faculty of Medicine, University of Oslo and Dept. of Gynaecology,, Oslo, Norway
- Dept of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Oppegaard KS, Qvigstad E, Fiala C, Heikinheimo O, Benson L, Gemzell-Danielsson K. Clinical follow-up compared with self-assessment of outcome after medical abortion: a multicentre, non-inferiority, randomised, controlled trial. Lancet. 2015 Feb 21;385(9969):698-704. doi: 10.1016/S0140-6736(14)61054-0. Epub 2014 Oct 30. PMID 25468164